CLINICAL TRIAL: NCT07336823
Title: A Clinical Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of JY232 Injection in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: JY232(JY232) Injection in Relapsed/Refractory Multiple Myeloma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shenzhen Genocury Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JY-CT-25-009
Record Dates: First submitted 2026-01-04; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A single-center, open-label, single-arm study of JY232 Injection (Experimental): This is a single-center, open-label, single-arm study to evaluate the efficacy and safety of intravenous JY232 Injection in patients with relapsed/refractory multiple myeloma. JY232 is designed to generate functional CAR-T cells directly within the body.
  Interventions: Drug: JY232 Injection

INTERVENTIONS:
Drug: JY232 Injection — This open-label, single-arm study is designed to evaluate the efficacy and safety of an in vivo Chimeric Antigen Receptor T-cell (CAR-T) therapy (JY232 preparation) in patients with relapsed or refractory multiple myeloma. Enrolled subjects will receive a single intravenous infusion of JY232, followed by a mandatory one-month in-hospital observation period for initial safety and efficacy assessments. Subsequently, subjects will enter a follow-up phase lasting up to 2 years to monitor long-term disease control.
  Other Names: in vivo CAR-T

SUMMARY:
This study is an investigator-initiated single center, single arm clinical study with a target population of patients with relapsed/refractory multiple myeloma. It is an early exploratory clinical study of the safety, tolerability and initial efficacy of JY232 injection in the treatment of relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
This open-label, single-arm study is designed to evaluate the efficacy and safety of in vivo CAR-T cell therapy (JY232 Injection) in patients with relapsed/refractory multiple myeloma. Following screening, eligible subjects will provide informed consent and be enrolled in the study. They will then receive JY232 Injection via intravenous infusion. Subsequently, subjects will undergo safety and efficacy assessments for up to 24 months to evaluate disease control.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily signs the informed consent form, is willing and able to comply with all study requirements.
2. Age 18-75 years, male or female.
3. Diagnosis of active MM according to the diagnostic criteria established by the International Myeloma Working Group (IMWG).
4. Must have undergone stem cell transplantation (SCT) or be transplant-ineligible.
5. Must have received at least 2 prior lines of anti-MM therapy (including immunomodulatory drugs, proteasome inhibitors, and anti-Cluster of Differentiation 38 (CD38) therapy, as single agents or in combination. Patients who are intolerant or have contraindications to these therapies are eligible for enrollment if they meet other inclusion/exclusion criteria). Each line of therapy must have included at least one complete cycle, and there must be documented evidence of disease progression on or relapse after the last line of therapy, or permanent discontinuation of therapy due to treatment-related toxicities (the reason for permanent discontinuation due to toxicity must be documented in the CRF). Furthermore, the patient must be refractory or intolerant to any established standard-of-care regimen that, in the investigator's assessment, is of significant clinical benefit to the patient.
6. The subject's tumor sample (bone marrow) tests positive for B-Cell Maturation Antigen (BCMA) expression on the plasma cell membrane via immunohistochemistry (IHC) or flow cytometry.
7. Presence of measurable disease at screening determined by any one of the following criteria:

   * Proportion of clonal plasma cells in bone marrow cytology, bone marrow biopsy histology, or flow cytometry ≥ 5%;
   * Serum monoclonal protein (M-protein) level: Immunoglobulin G (IgG) type M-protein ≥10 g/L; or Immunoglobulin A (IgA), Immunoglobulin D (IgD), Immunoglobulin E (IgE), Immunoglobulin M (IgM) type M-protein ≥5 g/L;
   * Urine M-protein level ≥200 mg/24 hours;
   * For MM without measurable serum or urine M-protein: involved serum free light chain ≥100 mg/L (10 mg/dL) and abnormal serum κ/λ free light chain ratio (<0.26 or >1.65);
   * Or clinical relapse: a. New bone lesions or soft tissue plasmacytomas (excluding osteoporotic fractures); b. Confirmed increase in Sum of the Product of Diameters (SPD) of existing plasmacytomas or bone lesions (≥50% increase in SPD of measurable lesions, absolute increase ≥1 cm).
8. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2 (see Appendix 1 for ECOG scale).
9. Expected survival time ≥12 weeks.
10. The subject must have adequate organ function, meeting all the following laboratory results prior to enrollment:

    * Hematology: Absolute neutrophil count (ANC) ≥ 1×10^9 /L (growth factor support is allowed, but must not have been administered within 7 days prior to the laboratory test); Absolute lymphocyte count (ALC) ≥0.3×10^9 /L; Platelets ≥50×10^9 /L (must not have received transfusion support within 7 days prior to the laboratory test); Hemoglobin ≥60 g/L (no red blood cell (RBC) transfusion within 7 days prior to the laboratory test; recombinant human erythropoietin is allowed);
    * Liver function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × upper limit of normal (ULN); Serum total bilirubin ≤1.5 × ULN;
    * Renal function: If available, measured CrCl from 24-hour urine collection; otherwise, calculated creatinine clearance (CrCl) via Cockcroft-Gault formula ≥ 40 ml/min;
    * Coagulation: Fibrinogen ≥1.0 g/L; Activated partial thromboplastin time (aPTT) ≤1.5 × ULN; Prothrombin time (PT) ≤1.5 × ULN;
    * Oxygen saturation >91% (on room air);
    * Left ventricular ejection fraction (LVEF) ≥ 50 %;
    * No clinically significant pericardial effusion detected.
11. The subject and their spouse agree to use effective barrier or pharmacological contraception from signing the informed consent until one year after CAR-T cell infusion (excluding the rhythm method).

Exclusion Criteria:

1. History of graft-versus-host disease (GvHD), or presence of autoimmune disease, immunodeficiency, or any condition requiring long-term immunosuppressive therapy.
2. Allogeneic hematopoietic stem cell transplantation within 6 months prior to infusion, or autologous hematopoietic stem cell transplantation within 3 months prior to infusion.
3. Prior anti-tumor therapy as follows:

   * Monoclonal antibody therapy for multiple myeloma (MM) within 21 days prior to dosing or within at least 5 half-lives (whichever is longer), or
   * Cytotoxic chemotherapy within 14 days prior to dosing or within at least 5 half-lives (whichever is longer), or
   * Proteasome inhibitor or immunomodulatory agent therapy within 14 days prior to dosing or within at least 5 half-lives (whichever is longer), or
   * Treatment with investigational drugs within 30 days prior to screening or within 5 half-lives (whichever is longer), or still within the washout period; or treatment involving invasive investigational medical devices, or
   * Radiotherapy within 4 weeks prior to dosing, or
   * Other anti-tumor therapies not listed above within 14 days prior to dosing or within at least 5 half-lives (whichever is longer).
4. Use of therapeutic doses of corticosteroids (defined as prednisone or equivalent > 20mg/day) within 7 days prior to screening, except for physiological replacement, topical, and inhaled steroids.
5. Hypertension uncontrolled by two or more antihypertensive medications to the following range (systolic BP <160 mmHg, diastolic BP <90 mmHg); or hypotension below normal range despite treatment (systolic BP <90 mmHg or diastolic BP <60 mmHg).
6. Severe cardiac disease: including but not limited to unstable angina, myocardial infarction (within 6 months prior to screening), congestive heart failure New York Heart Association (NYHA) class ≥III, severe arrhythmia.
7. Unstable systemic diseases as judged by the investigator: including but not limited to severe hepatic, renal, respiratory, or metabolic diseases requiring medication.
8. Diagnosis of malignancy other than MM within 5 years prior to screening, except for adequately treated carcinoma in situ of the cervix, basal cell or squamous cell skin cancer, localized prostate cancer treated with radical surgery, ductal carcinoma in situ of the breast treated with radical surgery.
9. History of solid organ transplantation.
10. Presence of central nervous system (CNS) involvement, symptoms of CNS involvement (including cranial nerve lesions and extensive lesions or spinal cord compression), or CNS metastasis.
11. MM patients with extramedullary disease (except for those with a single para-medullary lesion with a maximum transverse diameter ≤3cm).
12. MM patients with concomitant plasma cell leukemia (peripheral blood plasma cell proportion ≥5%).
13. Major surgery within 2 weeks prior to dosing, or planned surgery within 2 weeks after study treatment (subjects scheduled for local anesthesia surgery may participate).
14. Treatment with other interventional investigational drugs within 1 month prior to signing the informed consent form (ICF).
15. Uncontrolled active infection within 7 days prior to dosing, e.g., positive blood culture ≤72 hours prior to infusion (except for <CTCAE Grade 2 genitourinary tract and upper respiratory tract infections), or infection requiring medication.
16. Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with detectable Hepatitis B Virus (HBV) DNA ≥1×10^3 copies/mL in peripheral blood; positive for hepatitis C virus (HCV) antibody with detectable HCV RNA in peripheral blood; positive for human immunodeficiency virus (HIV) antibody; positive for cytomegalovirus (CMV) DNA; positive for syphilis.
17. Pregnant or breastfeeding women.
18. Psychiatric illness, impaired consciousness, or central nervous system disorders.
19. Non-hematological toxicities from prior therapy have not recovered to baseline or ≤ Grade 1 (per NCI-CTCAE v5.0, except for alopecia and Grade 2 peripheral neuropathy).
20. Any other condition considered by the investigator to be unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Related adverse events (AEs) | Up to 2 years after infusion
  The frequency, severity, and laboratory findings of all adverse events/serious adverse events are included.
Maximum Tolerated Dose (MTD) | Up to 28 days after infusion
  MTD will be determined based on Dose-Limiting Toxicities (DLTs ) observed during the first 28 days of study treatment.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 3 months after infusion
  Objective Response Rate (ORR) is defined as the proportion of subjects achieving stringent complete remission (sCR), complete remission (CR), very good partial response (VGPR) and partial response (PR).
Minimal Residual Disease (MRD) | Up to 3 months after infusion
  Flow cytometry-based MRD assessment, including the MRD-negative rate and duration of MRD negativity.
Best Overall Response | Up to 3 months after infusion
  The optimal degree of disease status improvement achieved by the patient over the course of the entire clinical trial or treatment period.
Duration of remission (DOR) | Up to 2 years after infusion
  Duration of remission (DOR) is the time from the first detection of CR or PR to the discovery of Progressive Disease (PD).
Time To Progression (TTP) | Up to 2 years after infusion
  The duration from the initiation of treatment until the first occurrence of objective disease progression.
Progression-free survival (PFS) | Up to 2 years after infusion
  Progression-free survival (PFS) is the time between the time a patient with tumor disease receives treatment and the time between the observation of disease progression or death from any cause.
Time to Complete Remission (TTCR) | Up to 2 years after infusion
  The time interval from the subject's receipt of JY232 treatment to the first documentation of a complete remission (CR) of the disease.
Overall survival (OS) | Up to 2 years after infusion
  Overall survival (OS) is the time from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ke Huang, Doctor, Study Chair — Shenzhen Genocury Biotech Co., Ltd.
Locations (1):
- Foshan First People's Hospital, Foshan, Guangdong, China

IPD SHARING:
Plan to Share IPD: No